CLINICAL TRIAL: NCT01736072
Title: RObotic Versus LAparoscopic Resection for Rectal Cancer An International, Multicentre, Prospective, Randomised, Controlled, Unblinded, Parallel-group Trial of Robotic-assisted Versus Laparoscopic Surgery for Treatment of Rectal Cancer.
Brief Title: RObotic Versus LAparoscopic Resection for Rectal Cancer
Acronym: ROLARR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: University of Leeds (Other)
Responsible Party: Principal Investigator, Nihn Tuan Nguyen, Professor and Interim Chair of Surgery, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20118537
Record Dates: First submitted 2012-11-15; First posted 2012-11-29 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; Colorectal Cancer; Laparoscopic Surgery; Robotic Surgery; Robotic Assisted Laparoscopic Surgery
MeSH Terms: conditions — Rectal Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic Resection of Rectal Cancer (Active Comparator): Research Subjects will be randomized to Surgical Resection of Rectal Cancer by Standard Laparoscopic Surgery.
  Interventions: Procedure: Standard Laparoscopic Surgery
- Robotic Resection of Rectal Cancer (Active Comparator): Research Subjects will be randomized to Surgical Resection of Rectal Cancer by Robotic Assisted Laparoscopic Surgery.
  Interventions: Procedure: Robotic Assisted Laparoscopic Surgery

INTERVENTIONS:
Procedure: Standard Laparoscopic Surgery — The research subjects will be randomized to Standard Laparoscopic Surgical procedure to resect their Rectal Cancer.
  Other Names: Laparoscopic Rectal Cancer Resection; Laparoscopic Cancer Resection; Rectal Cancer Surgery
  Arms: Laparoscopic Resection of Rectal Cancer
Procedure: Robotic Assisted Laparoscopic Surgery — The research subjects will be randomized Robotic Assisted Laparoscopic Surgical procedure to resect their Rectal Cancer.
  Other Names: Robotic Cancer Resection; Robotic Assisted Laparoscopic Rectal Cancer Resection; da Vinci Robotic System; Rectal Cancer Surgery
  Arms: Robotic Resection of Rectal Cancer

SUMMARY:
The purpose of this study is to compare two different surgical procedures for the treatment of Rectal Cancer: Laparoscopic Surgery and Robotic Assisted Laparoscopic Surgery. The ROLARR study is for participants with cancer of the rectum for whom a laparoscopic operation (sometimes called "keyhole surgery") has been recommended by their surgeon.

In the past most rectal cancers were removed using "open" surgery. Open surgery involves a large cut down the middle of the patient's abdomen to allow the surgeon to see and take out the cancer. On a previous study showed that using laparoscopic surgery to remove colorectal cancers was as good as open surgery for curing cancer.

There is now another option to remove rectal cancers, which involves using a robotic system with laparoscopic surgery. This type of surgery is called "robotic-assisted" laparoscopic surgery and is now becoming widely used by surgeons to remove cancers including the rectum, as well as for other non-cancer operations.

In order to perform robotic-assisted laparoscopic surgery, the surgeon sits at a robotic control unit a few feet away from the patient. Using the robotic control unit, the surgeon can see a clear video image of the patient's abdomen and the operation site. The surgeon can perform the operation from the robotic control unit by controlling the movement of a set of robotic surgical instruments, guided by the video camera.

Like standard laparoscopic surgery, the surgeon is able to carry out the entire operation through a few small cuts in the abdomen. The camera of the robotic system provides a 3D high-definition magnified view of the operation site and the robotic system is also able to translate the movements of the surgeon's hands into small precise movements inside the patient's body.

We want to test whether robotic-assisted laparoscopic surgery is as good, or even better, at removing rectal cancers as standard laparoscopic surgery (actually Robotic-assisted laparoscopic surgery is used as standard of care in rectal cancer patients at University of California, Irvine Medical Center). We also want to investigate whether using robotic-assisted laparoscopic surgery reduces the number of times a laparoscopic operation needs to be converted to an open operation, and see whether using a robotic system can also shorten the length of time patients need to stay in hospital and if it reduces the number of complications patients may have during and after their operation.

DETAILED DESCRIPTION:
The feasibility and safety of laparoscopic surgery has been established for colon cancer. The case for rectal cancer is less clear, and of the reported multicentre trials only the Medical Research Council (MRC) CLASICC trial included an evaluation of laparoscopic compared to open rectal cancer surgery. Although both laparoscopic and open rectal cancer resection were associated with similar lymph node yields, concern was expressed at the higher rate of circumferential resection margin (CRM) involvement in the laparoscopic arm (12.4%) as compared to the open arm (6.3%) for patients undergoing anterior resection. This however did not translate into a difference in local recurrence at either 3-year or 5-year follow-up. The difference in CRM involvement was felt to reflect the increased technical difficulties associated with the laparoscopic technique in the rectal cancer subgroup. This was supported by the higher conversion rate in the laparoscopic rectal subgroup (34%) as compared to the laparoscopic colon subgroup (25%). Analysis of CLASICC data revealed higher morbidity and mortality rates associated with laparoscopic cases converted to open operation (30-day morbidity: laparoscopic 29%, converted 45%; in-hospital mortality: laparoscopic 1%, converted 9%). Some of this increased morbidity may be related to more advanced cancers requiring conversion, but a proportion will inevitably have resulted from the increased operative time, increased technical difficulty, and the need for a laparotomy wound in converted cases.

The introduction of robotic-assisted laparoscopic surgery using the da Vinci™ system (Intuitive Surgical, California, USA) promises to eliminate many of the technical difficulties inherent in laparoscopic surgery. It offers the advantages of intuitive manipulation of laparoscopic instruments with 7-degrees of freedom of movement, a 3-dimensional field of view, a stable camera platform with zoom magnification, dexterity enhancement, and an ergonomic operating environment. Experience has shown that the benefits of the robot are most appreciated when surgical accuracy is required within a confined space, such as the pelvis.

Laparoscopic rectal cancer surgery is technically demanding requiring accurate pelvic dissection according to total mesorectal excision (TME) principles with autonomic nerve preservation. Inadvertent injury to the nerves has been attributed to the higher rate of male sexual dysfunction following laparoscopic surgery. The practicalities of robotic-assisted colorectal cancer surgery have been reported in small series but only two studies have concentrated on rectal cancer, and only one of these performed a randomised comparison in a small number of patients.

The literature on robotic-assisted colon surgery is limited to 17 small case series. Most of these comprise mixed benign and malignant disease. The largest by D'Annibale et al reported 53 robotic-assisted colectomies and compared outcomes with 53 laparoscopic resections. It concluded that robotic-assisted surgery was as safe and effective as laparoscopic, was particularly useful in pelvic dissection, but that cost-effectiveness needed further evaluation. Other reports concur that robotic-assisted colorectal surgery is feasible and safe, with low rates of conversion, morbidity and mortality, but with increased operative times. There is only one study which has addressed the issue of hospital costs. This compared 30 robotic-assisted with 27 standard laparoscopic cases and concluded that the total hospital cost was higher for robotic surgery.

The feasibility of robotics for TME rectal cancer resection was established by Pigazzi et al in a series of 6 low rectal cancers. A subsequent follow-up study of 39 rectal cancers treated prospectively by robotic-assisted resection reported a zero rate of conversion with a mortality of 0% and morbidity of 12.8%. The only randomised trial compared 18 patients assigned to robotic-assisted resection with 18 patients assigned to standard laparoscopic resection. No difference was observed in the operative times, the conversion rates (2 laparoscopic, 0 robotic), or the quality of mesorectal resection. The only difference was the length of hospital stay, which was significantly shorter following robotic-assisted laparoscopic surgery (robotic-assisted: 6.9 +/-1.3 days; standard laparoscopic: 8.7 +/-1.3 days, p<0.001) and attributed to a reduction in surgical trauma by the authors. In addition to original reports, there has been one systematic review of robotic-assisted colorectal surgery, which concluded that "robotic colorectal surgery is a promising field and may provide a powerful additional tool for optimal management of more challenging pathology, including rectal cancer".

The current proposal aims to test the hypothesis that robotic-assistance facilitates laparoscopic rectal cancer surgery. On short-term follow-up this should result in a reduction in the conversion rate and no worsening of the CRM positivity rate. On longer-term follow-up, the increased accuracy should improve post-operative bladder and sexual function, enhance quality of life (QoL), and ensure there is no increase in local disease recurrence.

There is a growing enthusiasm for robotics in many surgical specialities. This enthusiasm is often not supported by data on clinical or cost-effectiveness derived from rigorous evaluation by randomised controlled trials. This is the case for robotic-assisted rectal cancer surgery. Given the expense associated with the robotic systems and the limited evidence to support clinical and economic benefits, it is essential that a proper assessment of this new technology is performed in timely manner before its widespread recommendation or implementation. A randomized trial of robotic-assisted versus standard laparoscopic rectal cancer surgery is now urgently needed.

Rationale for current study

The safety and efficacy of robotic-assisted laparoscopic surgery have been established for certain operations, most notably radical prostatectomy. Pelvic surgery, including rectal cancer surgery, lends itself to robotic-assistance. However, the experience with robotic- assisted rectal cancer surgery is limited to a few small personal series and one randomised clinical trial. Although this data suggests it is feasible, it has not established a benefit over standard laparoscopic surgery in terms of technical, functional or oncological outcomes. The primary aim of any curative cancer surgery is complete oncological resection of the tumor with minimal morbidity. It is therefore of utmost importance that prior to the widespread use of robotics in rectal cancer surgery, it is subjected to rigorous evaluation. The use of this new technology incurs additional financial burdens on already overstretched health care resources and it is therefore essential to assess the health economics and cost- effectiveness in comparison to alternative treatments. As this trial is unlikely to be repeated, 3-year outcomes and cost effectiveness will be included within this trial. Specifically, it is aimed to provide information on the ability of the robotic system to facilitate laparoscopic rectal cancer resection, its impact on oncological outcomes (short-term and long-term), its effect on functional outcomes and QoL, and its cost-effectiveness in terms of future healthcare decision-making. Currently, and for the foreseeable future, there is only one surgical robotic system, the da Vinci™ robot. To avoid any criticism of commercial bias, it is imperative that an evaluation of this robotic technology is performed independently of the manufacturer.

Justification for a randomized controlled trial

Since this is a new technology, it is essential that a proper evaluation is performed and disseminated prior to its widespread implementation. A timely assessment is imperative and for this reason there is no plan to perform a prior pilot study, which would inevitably delay evaluation by proper scientific methods. The feasibility of robotic-assisted rectal cancer surgery has already been established and preliminary data upon which to base sample size calculations are available. The time is right for a formal randomised controlled trial to provide a definitive answer to the proposed research question.

Aims and Objectives

The purpose of the trial is to perform a rigorous evaluation of robotic-assisted rectal cancer surgery by means of a randomised, controlled trial. The chosen comparator is standard laparoscopic rectal cancer resection, which is essentially the same procedure but without the use of the robotic device. The two operative interventions will be evaluated for short- and longer-term outcomes. The key short-term outcomes will include assessment of technical ease of the operation, as determined by the clinical indicator of low conversion rate to open operation, and clear pathological resection margins as an indicator of surgical accuracy and improved oncological outcome. In addition, QoL assessment and analysis of cost- effectiveness will be performed to aid evidence-based knowledge to inform National Health Service (NHS) and other service providers and decision-makers. These short-term outcomes will be analyzed after the last randomised patient has had 6 months of follow-up to provide a timely assessment of the new technology, and made available to the public, clinicians and healthcare providers to inform health-care decision making. Longer-term outcomes will concentrate on oncological aspects of the disease and its surgical treatment with analysis of disease-free and overall survival and local recurrence rates at 3-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years
2. Able to provide written informed consent
3. Diagnosis of rectal cancer amenable to curative surgery either by low anterior resection, high anterior resection, or abdominoperineal resection i.e. staged T1-3, N0-2, M0 by imaging as per local practice; although not mandated, CT imaging with either additional MRI or trans-rectal ultrasound is recommended to assess distant and local disease.
4. Rectal cancer suitable for resection by either standard or robotic-assisted laparoscopic procedure
5. Fit for robotic-assisted or standard laparoscopic rectal resection
6. American Society of Anesthesiologists (ASA) physical status ≤ 3
7. Capable of completing required questionnaires at time of consent (provided questionnaires are available in a language spoke fluently by the participant)

Exclusion Criteria:

1. Benign lesions of the rectum
2. Benign or malignant diseases of the anal canal
3. Locally advanced cancers not amenable to curative surgery
4. Locally advanced cancers requiring en bloc multi-visceral resection
5. Synchronous colorectal tumors requiring multi-segment surgical resection (N.B. a benign lesion within the resection field in addition to the main cancer would not exclude a patient)
6. Co-existent inflammatory bowel disease
7. Clinical or radiological evidence of metastatic spread
8. Concurrent or previous diagnosis of invasive cancer within 5 years that could confuse diagnosis (non- melanomatous skin cancer or superficial bladder cancer treated with curative intent are acceptable; for other cases please discuss with Chief Investigator via CTRU)
9. History of psychiatric or addictive disorder or other medical condition that, in the opinion of the investigator, would preclude the patient from meeting the trial requirements
10. Pregnancy or breastfeeding women.
11. Participation in another rectal cancer clinical trial relating to surgical technique.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 471 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
End of Conversion to Open Surgery | 1 day
  The primary end point is the rate of conversion to open surgery as an indicator of surgical technical difficulty. Conversion is defined as the use of a laparotomy wound for any part of the mesorectal dissection. The use of a limited laparotomy wound to facilitate a low stapled anastomosis and/or specimen extraction is permissible and not defined as an open conversion.

SECONDARY OUTCOMES:
Oncological Efficacy | 1 day
  Pathological CRM positivity rates as recorded from local histopathology review, where resection margin positivity is defined as a distance of ≤1mm of the cancer from any resection margin.

OTHER OUTCOMES:
Intra-operative and post-operative complications | 30 day and 6 months
  All the intra-operative complications will be assessed at 30 days and 6-months after the surgical procedure.
30-day post-operative Mortality | 30 day post-surgery
  Thirty-day operative mortality is defined as deaths occurring from any cause during the first 30 post-operative days.
Three-year disease-free and overall survival. | 3 years
  Overall survival is defined as the time from date of randomization to date of death from any cause. Disease-free survival is defined according to Punt et al's definitions as the time from date of randomization to date of death from any cause, recurrent disease (locoregional or distant recurrence) or second primary cancer.
Sexual Disfunction Assessment | 6-months
  Patient self-reported bladder and sexual function as assessed by the International Prostatic Symptom Score(I-PSS©) for male and female bladder function, and the International Index of Erectile Function (IIEF) Female Sexual Function Index(FSFI©) for sexual function.

CONTACTS AND LOCATIONS:
Overall Officials: Alessio Pigazzi, MD, Principal Investigator — University of California, Irvine
Locations (8):
- United States (8):
  - John Muir Medical Center, Concord, California
  - University of California, Irvine Medical Center, Orange, California
  - Jackson South Community Hospital, Miami, Florida
  - St. Joseph Mercy Health System, Ypsilanti, Michigan
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Aria Health, Philadelphia, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jayne DG, Guillou PJ, Thorpe H, Quirke P, Copeland J, Smith AM, Heath RM, Brown JM; UK MRC CLASICC Trial Group. Randomized trial of laparoscopic-assisted resection of colorectal carcinoma: 3-year results of the UK MRC CLASICC Trial Group. J Clin Oncol. 2007 Jul 20;25(21):3061-8. doi: 10.1200/JCO.2006.09.7758. PMID 17634484
- [Background] Clinical Outcomes of Surgical Therapy Study Group; Nelson H, Sargent DJ, Wieand HS, Fleshman J, Anvari M, Stryker SJ, Beart RW Jr, Hellinger M, Flanagan R Jr, Peters W, Ota D. A comparison of laparoscopically assisted and open colectomy for colon cancer. N Engl J Med. 2004 May 13;350(20):2050-9. doi: 10.1056/NEJMoa032651. PMID 15141043
- [Background] Tang CL, Eu KW, Tai BC, Soh JG, MacHin D, Seow-Choen F. Randomized clinical trial of the effect of open versus laparoscopically assisted colectomy on systemic immunity in patients with colorectal cancer. Br J Surg. 2001 Jun;88(6):801-7. doi: 10.1046/j.1365-2168.2001.01781.x. PMID 11412248
- [Background] Guillou PJ, Quirke P, Thorpe H, Walker J, Jayne DG, Smith AM, Heath RM, Brown JM; MRC CLASICC trial group. Short-term endpoints of conventional versus laparoscopic-assisted surgery in patients with colorectal cancer (MRC CLASICC trial): multicentre, randomised controlled trial. Lancet. 2005 May 14-20;365(9472):1718-26. doi: 10.1016/S0140-6736(05)66545-2. PMID 15894098
- [Background] Taylor GW. Minimally Invasive Robotic Association 2nd international congress: the Union League Club, New York, NY, USA, 18-20 January 2007. Int J Med Robot. 2007 Sep;3(3):281-6. doi: 10.1002/rcs.154. PMID 17924452
- [Background] Jayne DG, Brown JM, Thorpe H, Walker J, Quirke P, Guillou PJ. Bladder and sexual function following resection for rectal cancer in a randomized clinical trial of laparoscopic versus open technique. Br J Surg. 2005 Sep;92(9):1124-32. doi: 10.1002/bjs.4989. PMID 15997446
- [Background] Hildebrandt U, Plusczyk T, Kessler K, Menger MD. Single-surgeon surgery in laparoscopic colonic resection. Dis Colon Rectum. 2003 Dec;46(12):1640-5. doi: 10.1007/BF02660769. PMID 14668589
- [Background] DeNoto G, Rubach E, Ravikumar TS. A standardized technique for robotically performed sigmoid colectomy. J Laparoendosc Adv Surg Tech A. 2006 Dec;16(6):551-6. doi: 10.1089/lap.2006.16.551. PMID 17243868
- [Background] Baik SH, Ko YT, Kang CM, Lee WJ, Kim NK, Sohn SK, Chi HS, Cho CH. Robotic tumor-specific mesorectal excision of rectal cancer: short-term outcome of a pilot randomized trial. Surg Endosc. 2008 Jul;22(7):1601-8. doi: 10.1007/s00464-008-9752-z. Epub 2008 Feb 13. PMID 18270772
- [Background] Pigazzi A, Ellenhorn JD, Ballantyne GH, Paz IB. Robotic-assisted laparoscopic low anterior resection with total mesorectal excision for rectal cancer. Surg Endosc. 2006 Oct;20(10):1521-5. doi: 10.1007/s00464-005-0855-5. Epub 2006 Aug 1. PMID 16897284
- [Background] D'Annibale A, Morpurgo E, Fiscon V, Trevisan P, Sovernigo G, Orsini C, Guidolin D. Robotic and laparoscopic surgery for treatment of colorectal diseases. Dis Colon Rectum. 2004 Dec;47(12):2162-8. doi: 10.1007/s10350-004-0711-z. PMID 15657669
- [Background] Rawlings AL, Woodland JH, Crawford DL. Telerobotic surgery for right and sigmoid colectomies: 30 consecutive cases. Surg Endosc. 2006 Nov;20(11):1713-8. doi: 10.1007/s00464-005-0771-8. Epub 2006 Aug 28. PMID 17008953
- [Background] Rawlings AL, Woodland JH, Vegunta RK, Crawford DL. Robotic versus laparoscopic colectomy. Surg Endosc. 2007 Oct;21(10):1701-8. doi: 10.1007/s00464-007-9231-y. Epub 2007 Mar 13. PMID 17353988
- [Background] Hellan M, Anderson C, Ellenhorn JD, Paz B, Pigazzi A. Short-term outcomes after robotic-assisted total mesorectal excision for rectal cancer. Ann Surg Oncol. 2007 Nov;14(11):3168-73. doi: 10.1245/s10434-007-9544-z. Epub 2007 Sep 1. PMID 17763911
- [Background] Mirnezami AH, Mirnezami R, Venkatasubramaniam AK, Chandrakumaran K, Cecil TD, Moran BJ. Robotic colorectal surgery: hype or new hope? A systematic review of robotics in colorectal surgery. Colorectal Dis. 2010 Nov;12(11):1084-93. doi: 10.1111/j.1463-1318.2009.01999.x. PMID 19594601
- [Background] Vassiliou MC, Feldman LS, Andrew CG, Bergman S, Leffondre K, Stanbridge D, Fried GM. A global assessment tool for evaluation of intraoperative laparoscopic skills. Am J Surg. 2005 Jul;190(1):107-13. doi: 10.1016/j.amjsurg.2005.04.004. PMID 15972181
- [Background] Barry MJ, Fowler FJ Jr, O'Leary MP, Bruskewitz RC, Holtgrewe HL, Mebust WK, Cockett AT. The American Urological Association symptom index for benign prostatic hyperplasia. The Measurement Committee of the American Urological Association. J Urol. 1992 Nov;148(5):1549-57; discussion 1564. doi: 10.1016/s0022-5347(17)36966-5. PMID 1279218
- [Background] Rosen RC, Riley A, Wagner G, Osterloh IH, Kirkpatrick J, Mishra A. The international index of erectile function (IIEF): a multidimensional scale for assessment of erectile dysfunction. Urology. 1997 Jun;49(6):822-30. doi: 10.1016/s0090-4295(97)00238-0. PMID 9187685
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Smets EM, Garssen B, Cull A, de Haes JC. Application of the multidimensional fatigue inventory (MFI-20) in cancer patients receiving radiotherapy. Br J Cancer. 1996 Jan;73(2):241-5. doi: 10.1038/bjc.1996.42. PMID 8546913
- [Background] Sobin LH, Fleming ID. TNM Classification of Malignant Tumors, fifth edition (1997). Union Internationale Contre le Cancer and the American Joint Committee on Cancer. Cancer. 1997 Nov 1;80(9):1803-4. doi: 10.1002/(sici)1097-0142(19971101)80:93.0.co;2-9. No abstract available. PMID 9351551
- [Background] Punt CJ, Buyse M, Kohne CH, Hohenberger P, Labianca R, Schmoll HJ, Pahlman L, Sobrero A, Douillard JY. Endpoints in adjuvant treatment trials: a systematic review of the literature in colon cancer and proposed definitions for future trials. J Natl Cancer Inst. 2007 Jul 4;99(13):998-1003. doi: 10.1093/jnci/djm024. Epub 2007 Jun 27. PMID 17596575
- [Background] Aziz O, Constantinides V, Tekkis PP, Athanasiou T, Purkayastha S, Paraskeva P, Darzi AW, Heriot AG. Laparoscopic versus open surgery for rectal cancer: a meta-analysis. Ann Surg Oncol. 2006 Mar;13(3):413-24. doi: 10.1245/ASO.2006.05.045. Epub 2006 Feb 1. PMID 16450220
- [Background] Moloo H, Mamazza J, Poulin EC, Burpee SE, Bendavid Y, Klein L, Gregoire R, Schlachta CM. Laparoscopic resections for colorectal cancer: does conversion survival? Surg Endosc. 2004 May;18(5):732-5. doi: 10.1007/s00464-003-8923-1. Epub 2004 Apr 6. PMID 15216851
- [Background] Wibe A, Syse A, Andersen E, Tretli S, Myrvold HE, Soreide O; Norwegian Rectal Cancer Group. Oncological outcomes after total mesorectal excision for cure for cancer of the lower rectum: anterior vs. abdominoperineal resection. Dis Colon Rectum. 2004 Jan;47(1):48-58. doi: 10.1007/s10350-003-0012-y. Epub 2004 Jan 14. PMID 14719151
- [Background] Shepherd NA, Baxter KJ, Love SB. Influence of local peritoneal involvement on pelvic recurrence and prognosis in rectal cancer. J Clin Pathol. 1995 Sep;48(9):849-55. doi: 10.1136/jcp.48.9.849. PMID 7490320
- [Background] Dworak O, Keilholz L, Hoffmann A. Pathological features of rectal cancer after preoperative radiochemotherapy. Int J Colorectal Dis. 1997;12(1):19-23. doi: 10.1007/s003840050072. PMID 9112145
- See also: ROLARR Trial CTRU University of Leeds — http://medhealth.leeds.ac.uk/news/article/182/rolarr_trial_update